CLINICAL TRIAL: NCT05011162
Title: "REACT-FM" Real-World Evidence From Smartphone-Based Acceptance and Commitment Therapy in Fibromyalgia
Acronym: REACT-FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swing-003
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a virtual, single-arm, pragmatic, non-significant risk study.
  Study participants will receive 12 weeks of Digital Acceptance and Commitment Therapy (ACT) in addition to their standard care for fibromyalgia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Digital Acceptance and Commitment Therapy (ACT) Arm (Other): Pragmatic
  Interventions: Device: Digital ACT

INTERVENTIONS:
Device: Digital ACT — Study participants will receive 12 weeks of Digital Acceptance and Commitment Therapy (ACT).

SUMMARY:
The objective of this study is to assess the clinical impact of a digital therapy for the management of fibromyalgia. Study participants receive 12 weeks of Digital Acceptance and Commitment Therapy (ACT) in addition to their standard care for fibromyalgia. The primary endpoint is the Patient Global Impression of Change (PGIC) at week 12. This is a virtual, single-arm, pragmatic, non-significant risk study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant is 22 years of age or older
2. Participant has a diagnosis of fibromyalgia based on self-reported responses to 2016 ACR criteria for fibromyalgia diagnosis
3. Participant is capable of reading and understanding English and has provided written informed consent to participate (signed electronically).

Key Exclusion Criteria:

1. Participant is not a resident of the United States
2. In the opinion of the Investigator or Sponsor, the participant suffers from a severe psychiatric condition
3. Participant has a diagnosis of, or is being treated for any type of Dementia (Parkinson's disease, Alzheimer's Disease, Huntington's Disease, Lewy Body Dementia, Creuztfeldt-Jacob Disease, Frontotemporal Dementia, Korsakoff Syndrome, Vascular Dementia) or a current diagnosis of cancer or recurrence in the past 3 years (other than basal or squamous cell skin cancer)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) Response | Week 12
  PGIC scores included are: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score | Baseline to Week 12
  FIQ-R total score ranges between 0-100 with a reduction in score indicating reduced fibromyalgia severity.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) impact domain score | Baseline to Week 12
  FIQ-R impact domain score ranges between 0-20 with a reduction in score indicating reduced fibromyalgia impact.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) symptoms domain score | Baseline to Week 12
  FIQ-R symptoms domain score ranges between 0-50 with a reduction in score indicating reduced fibromyalgia symptoms.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) function domain score | Baseline to Week 12
  FIQ-R function domain score ranges between 0-30 with a reduction in score indicating improved function.
Participant's self-reported average weekly pain score, recorded on an NRS scale | Baseline to Week 12
  Average pain intensity score ranges between 0-10 with a reduction in score indicating a decrease in pain intensity.
Participant's self-reported average weekly pain interference score, recorded on an NRS scale | Baseline to Week 12
  Average pain interference score ranges between 0-10 with a reduction in score indicating a decrease in pain interference.
Participant's self-reported weekly sleep interference score, recorded on an NRS scale | Baseline to Week 12
  Average sleep interference score ranges between 0-10 with a reduction in score indicating a decrease in sleep interference.
Participant's engagement with the Digital ACT device | Weeks 1-12
  Participant engagement will be assessed by evaluating the following:
  Average days engaged in treatment per week (number of days opening the device), with a higher score indicating more engagement.
Participant's engagement with the Digital ACT device | Weeks 1-12
  Participant engagement will be assessed by evaluating the following:
  Average number of completed sessions per week, with a higher score indicating more engagement.
Participant's compliance with the Digital ACT device | Weeks 1-12
  Participant compliance will be assessed by evaluating the percentage of participants who completed the core program within the study time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keefe, MD, Principal Investigator — Swing Therapeutics
Locations (1):
- Swing Therapeutics, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Swing Therapeutics Website — https://www.swingtherapeutics.com/